CLINICAL TRIAL: NCT00785811
Title: Randomized, Double Blind, Placebo Controlled Study of Parallel Groups to Evaluate the Effect of Chronic Supplementation of L-arginine in the Muscular Performance.
Brief Title: Effect of Chronic Supplementation of L-arginine in the Muscular Performance
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Required by the investigator. The site could not recruit patients anymore.
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: LARAS_L_02921
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2011-03-16 (Estimated); Status verified 2011-03

CONDITIONS: Muscular Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): L-arginine aspartate (Targifor)
  Interventions: Drug: L-arginine aspartate (Targifor)
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo L-arginine aspartate (Targifor)

INTERVENTIONS:
Drug: L-arginine aspartate (Targifor) — 3g of L-arginine taken orally in a single daily dose for 8 weeks
  Arms: 1
Drug: Placebo L-arginine aspartate (Targifor) — Placebo of L-arginine taken orally in a single daily dose for 8 weeks
  Arms: 2

SUMMARY:
The primary purpose of this study is to evaluate the effect of oral administration of L-arginine in the muscular fatigue of the quadriceps, expressed in terms of the Fatigue Resistance Factor (FRF). The secondary purpose of this study is to evaluate the effect of oral administration of L-arginine in the muscular force the quadriceps.

ELIGIBILITY:
Inclusion criteria:

Healthy young adults for both sex; Age between 20 and 55 years; Slight or moderate physical activity, 30 minutes per day, at least 3 times a week;

Exclusion criteria:

Cardiac or pulmonary disease; Previous history of knee surgery or skeletal muscular dysfunctions in hip, knee or ankle joints; Athletic person (intensive anaerobic activity); None practiced of physical activity regularly; Medications usage

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2008-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Fatigue Resistance Factor (FRF) | Throughout the study

SECONDARY OUTCOMES:
Maximum force in Newton (N) and fast or explosive force | at time 30% of the maximum isometric force
Maximum force in Newton (N) and fast or explosive force | at time 50% of the maximum isometric force
Maximum force in Newton (N) and fast or explosive force | at time 90% of the maximum isometric force

CONTACTS AND LOCATIONS:
Overall Officials: Jaderson Lima, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, São Paulo, Brazil